CLINICAL TRIAL: NCT06139744
Title: Efficacy and Safety of Dietary Supplementation of Diamine Oxidase (DAO) to Improve Symptoms in Patients With Irritable Bowel Syndrome
Brief Title: Efficacy and Safety of Dietary Supplementation of Diamine Oxidase to Improve Symptoms in Patients With IBS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Chief physician, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20230915-01
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAO supplement group (Experimental): One tablet of the supplementary study product was taken orally before morning, lunch and dinner every day, and each tablet contained 4.2mg of dehydrated pea seedling powder.
  Interventions: Drug: DAO supplement
- Placebo group (Placebo Comparator): Placebo was orally supplemented with one tablet each day before morning, lunch and dinner, and placebo did not contain dehydrated pea seedling powder 4.2mg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAO supplement — One tablet of the supplementary study product is taken orally before morning, lunch and dinner every day, and each tablet contains 4.2mg of dehydrated pea seedling powder.
  Other Names: PEA SPROUT DEHYDRATED POWDER
  Arms: DAO supplement group
Drug: Placebo — Placebo is orally supplemented with one tablet each day before morning, lunch and dinner, and placebo does not contain dehydrated pea seedling powder 4.2mg.
  Arms: Placebo group

SUMMARY:
This project is a single center, randomized, controlled clinical trial evaluating the effects of DAO enzyme dietary supplement on symptoms of irritable bowel syndrome.

These participants are randomized to either a 4-week group with DAO enzyme dietary supplement or placebo. The participants are required to fill out IBS-SSS and IBS-QOL questionnaires and record their IBS symptom improvement, IBS treatment drug use, compliance and adverse reactions every evening. At the same time, the patients' diet is continuously recorded for 3 days by 24-hour diet review method in Visit 0, Visit 1 and Visit 2, respectively, to inform the patients to avoid large fluctuations in diet structure. On days 0, 14 and 28, the subjects are asked to visit the hospital offline. The staff check with the subjects in detail according to the scale and questionnaire contents, and review the general situation and questionnaire in the previous 2 weeks. On the 7th and 21st day, the staff contact the subjects online to provide guidance and remind the subjects to fill in the scale and questionnaire. In addition, oral mucosal samples, urine and feces will be collected for identifying mutations in the genetic DAO enzyme coding gene, histamine detection and 16sRNA sequencing, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. Diagnosed with IBS according to Rome IV diagnostic criteria; Recurrent abdominal pain occurred on an average of at least 1 day per week in the past 3 months and was associated with two or more of the following criteria: i. Related to defecation; ii. Associated with changes in bowel frequency; iii. Correlated with fecal morphological changes. The symptoms appeared at least 6 months before diagnosis, and the above diagnostic criteria were met in the last 3 months.
3. Voluntarily participate in the experiment and sign the informed consent.

Exclusion Criteria:

1. Patients with endoscopy examinations which suggest chronic intestinal diseases other than IBS, such as inflammatory bowel disease, celiac disease, gastric and duodenal ulcers, parasitic or bacterial intestinal infections;
2. Pregnant and lactating women;
3. Patients suffering from serious concomitant diseases, such as liver disease, cardiovascular disease, lung disease, kidney disease, tumor;
4. Alcoholism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS | 4 weeks of study medication administration
  The effects of DAO enzyme dietary supplement from dehydrated pea seedling powder on IBS symptoms were evaluated by the Severity Scale of irritable bowel Syndrome (IBS-SSS) and the changes of several independent symptoms.

SECONDARY OUTCOMES:
IBS-QOL | 4 weeks of study medication administration
  The overall improvement of quality of life in IBS patients with DAO enzyme dietary supplement from dehydrated pea seedling powder was evaluated by the irritable bowel Syndrome Quality of Life Questionnaire (IBS-QOL).
Improvement of symptoms listed in the Rome IV diagnostic criteria for IBS | 4 weeks of study medication administration
  1. Number of days with abdominal pain in the past week;
  2. Number of days of defecation-related abdominal pain in the past week;
  3. Frequency of bowel movements;
  4. Changes in stool pattern according to the Bristol stool Classification Scale.

OTHER OUTCOMES:
Effect of diet difference on treatment of IBS with dehydrated pea seedling powder | 4 weeks of study medication administration
  The effects of dietary differences on the treatment of IBS with dehydrated pea seedling powder were evaluated by 24-hour diet review.
Histamine concentration in urine | 4 weeks of study medication administration
  The effect of dehydrated pea seedling powder on histamine concentration was evaluated by detecting histamine concentration in urine.
Fecal intestinal flora | 4 weeks of study medication administration
  Changes of fecal intestinal flora in patients before and after oral administration of dehydrated pea seedling powder
The expression of diamine oxidase in IBS patients | before study medication administration
  The expression of diamine oxidase in IBS patients
Drug use in subjects | 4 weeks of study medication administration
  The effects of dehydrated pea seedling powder interventions on drug use in subjects
Adverse events | 4 weeks of study medication administration
  The occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Zhenyu Zhang, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No